CLINICAL TRIAL: NCT04173273
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Study to Assess the Efficacy and Safety of Oral Etrasimod as Induction and Maintenance Therapy for Moderately to Severely Active Crohn's Disease
Brief Title: A Study Evaluating the Efficacy and Safety of Oral Etrasimod in the Treatment of Adult Participants With Moderately to Severely Active Crohn's Disease
Acronym: CULTIVATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to a lack of efficacy in sub-study 1
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD334-202; C5041006 (Other: Alias Study Number); NCT05033340 (obsolete NCT alias)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Crohn's Disease
Keywords: Etrasimod; Crohn's disease; APD334; Inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Etrasimod Dose A (Experimental)
  Interventions: Drug: Etrasimod
- Etrasimod Dose B (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Dose A taken by mouth, once daily.
  Other Names: APD334
  Arms: Etrasimod Dose A
Drug: Etrasimod — Dose B taken by mouth, once daily.
  Other Names: APD334
  Arms: Etrasimod Dose B
Drug: Placebo — Etrasimod matching placebo tablet taken by mouth, once daily.
  Arms: Placebo

SUMMARY:
This is a Phase 2/3 study that comprises 5 substudies designed to evaluate the efficacy, safety, and tolerability of oral etrasimod as therapy in adult participants with moderately to severely active Crohn's disease (CD) who are refractory or intolerant to at least 1 of the current therapies for CD (ie, corticosteroids, immunosuppressants, or biologics). The overall duration of this study is up to 282 weeks, inclusive of the Screening Period, Treatment Period of up to 274 weeks (Induction, Extension or Maintenance, and Long-term Extension Periods), and the 4-Week Follow-Up Period for safety assessment.

DETAILED DESCRIPTION:
This study includes 5 substudies:

Substudy A - Phase 2: A Phase 2, randomized, double-blind, substudy to assess the safety, tolerability, and efficacy of oral etrasimod therapy in participants with moderate to severe CD that supports the selection of an induction and maintenance dose(s) for Phase 3.

Substudy 1 - Phase 2: A Phase 2b randomized, double-blind, placebo-controlled, dose-ranging induction substudy to evaluate etrasimod as induction therapy and select an induction and maintenance dose(s) for continued evaluation in Phase 3.

Substudy 2 - Induction: A Phase 3 randomized, double-blind, placebo-controlled substudy to evaluate etrasimod as induction therapy.

Substudy 3 - Maintenance: A Phase 3 randomized, double-blind, placebo-controlled substudy to evaluate etrasimod as maintenance therapy. Participants from Substudy 1 and Substudy 2 will be enrolled in Substudy 3.

Substudy 4 - Long-Term Extension: A long-term extension substudy for participants who complete at least 52 weeks of treatment. Participants from Substudy 3 and Substudy A are planned to be enrolled in Substudy 4.

ELIGIBILITY:
Eligibility criteria applicable to all substudies:

Inclusion Criteria:

* Men or women 18 to 80 years of age,
* Ability to provide written informed consent or assent and to be compliant with the schedule of protocol assessments
* Diagnosed with Crohn's disease (CD) ≥ 3 months
* Have moderately to severely active CD at Screening
* Demonstrated inadequate response (ie, primary non-response), loss of response to, or intolerance to ≥ 1 of the following therapies for the treatment of CD:

  1. Oral corticosteroids (eg, prednisone or its equivalent, budesonide)
  2. Immunosuppressants (eg, azathioprine [AZA], 6 mercaptopurine [6-MP], or methotrexate [MTX])
  3. Tumor necrosis factor alpha (TNFα) antagonists (eg, infliximab, adalimumab, certolizumab pegol, or biosimilars)
  4. Integrin receptor antagonist (eg, vedolizumab)
  5. Interleukin -12/-23 antagonist (eg, ustekinumab)
* Females of childbearing potential must be nonpregnant
* Females of childbearing potential and males must use contraception

Exclusion Criteria:

* History of inadequate response (ie, primary non-response) to agents from ≥ 2 classes of biologics marketed for the treatment of CD (ie, TNFα antagonists, interleukin 12/ 23 antagonist, and integrin receptor antagonist).
* Have ulcerative colitis, indeterminate colitis, microscopic colitis, ischemic colitis, radiation colitis, diverticular disease associated colitis, toxic megacolon, or active infectious colitis or test positive for Clostridioides difficile toxin at Screening.
* Have functional or post-operative short-bowel syndrome or any associated complications that may require surgery or interfere with efficacy assessments
* Had surgical treatment for intra abdominal abscesses ≤ 8 weeks prior to randomization or surgical treatment for perianal abscesses ≤ 4 weeks prior to randomization.
* Had intestinal resection ≤ 24 weeks prior to randomization or other intra abdominal surgeries ≤ 12 weeks prior to randomization.
* Have an ileostomy or a colostomy.

Inclusion Criteria for Substudy 3:

- Participants who entered the Extended Induction Period of Substudy 1 and Substudy 2 must have completed the Extended Induction -Week 6 Visit

Inclusion Criteria for Substudy 4:

- Participant must have completed the Week 52 Visit of Substudy 3 or the Week 66 Visit of Substudy A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with Endoscopic Response [Substudy A] | Weeks 14 and 52
Proportion of Participants With Endoscopic Response [Substudy 1] | Week 14
Proportion of Participants With Endoscopic Response [Substudy 2] | Week 14
Proportion of Participants With Clinical Remission Crohn's Disease Activity Index (CDAI) [Substudy 2] | Week 14
Proportion of Participants With Clinical Remission CDAI [Substudy 3] | Week 52
Proportion of Participants With Endoscopic Response [Substudy 3] | Week 52

SECONDARY OUTCOMES:
Proportion of Participants With Clinical Remission CDAI [Substudy A] | Up to Week 66
Change From Baseline in Simple Endoscopic Score in Crohn's Disease (SES-CD) Score [Substudy A] | Baseline to Week 66
Change From Baseline in CDAI Score [Substudy A] | Baseline to Week 66
Proportion of Participants With Clinical Remission CDAI [Substudy 1] | Week 14
Proportion of Participants with Clinical Remission Patient Reported Outcome 2 (PRO2) [Substudy 1] | Week 14
Proportion of Participants With Clinical Remission Patient Reported Outcome 2 (PRO2) [Substudy 2] | Week 14
Proportion of Participants With Clinical Response CDAI [Substudy 2] | Week 14
Proportion of Participants With Endoscopic Response and Clinical Remission CDAI [Substudy 2] | Week 14
Proportion of Participants With Endoscopic Remission [Substudy 2] | Week 14
Change from baseline in CD-PRO/SS [Substudy 2] | Week 14
Proportion of Participants With Clinical Remission CDAI Among Participants In Clinical Remission CDAI at Substudy 3 Baseline [Substudy 3] | Week 52
Proportion of Participants With Endoscopic Response Among Participants in Endoscopic Response at Substudy 3 Baseline [Substudy 3] | Week 52
Proportion of Participants With Corticosteroid-Free Clinical Remission CDAI Among Participants Receiving Corticosteroids at Substudy 3 Baseline [Substudy 3] | Week 52
Proportion of Participants With Endoscopic Remission [Substudy 3] | Week 52
Proportion of Participants With Clinical Remission PRO2 [Substudy 3] | Week 52
Proportion of Participants with Clinical Response or Endoscopic Response [Substudy 3] | Week 52
Proportion of Participants With Clinical Remission CDAI by Visit up to the End Of Treatment [Substudy 4] | Up to Week 208
Proportion of Participants With Clinical Remission PRO2 by Visit up to the End Of Treatment [Substudy 4] | Up to Week 208
Number and Severity of Adverse Events | Up to approximately 70 weeks for Substudy A,approximately 24 weeks for Substudy 1 and 2; 42 weeks for Substudy 3; and 212 weeks for Substudy 4
  Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (518):
- United States (191):
  - Center for Digestive Health (Endoscopy Location), Dothan, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - Dothan Eyecare-Dr. Brent McKinley (OCT Location), Dothan, Alabama
  - Pulmonary Associates (PFT Location), Dothan, Alabama
  - Flowers Hospital (Imaging Location), Dothan, Alabama
  - Digestive Health Specialists (Satellite Clinic Location), Mobile, Alabama
  - Premier Medical Group East (Opthalmology & Optometry Facility), Mobile, Alabama
  - Pulmonary Associates (Chest X-Ray & PFT Facility), Mobile, Alabama
  - Surgicare of Mobile (Endoscopy & Biopsy Facility), Mobile, Alabama
  - Arizona Retina Institute/ Phoenix Retina Associates(OCT), Peoria, Arizona
  - SimonMed Imaging (Imaging), Peoria, Arizona
  - Sun City Endoscopy Center (Endoscopy), Sun City, Arizona
  - Om Research LLC, Apple Valley, California
  - Victor Valley Advanced Imaging, Apple Valley, California
  - Koman Family Outpatient Pavilion (ENDO), La Jolla, California
  - Perlman Medical Offices, La Jolla, California
  - UCSD Clinical and Translational Research Institute, La Jolla, California
  - UCSD Health System (Endo/PFT/DLCO), La Jolla, California
  - UCSD lnvestigational Drug Service Pharmacy, La Jolla, California
  - Shiley Eye Institute (OCT), La Jolla, California
  - A V Pediatrics, Allergy and Family Medicine - PFT, Lancaster, California
  - Advanced Endoscopy and Pain Center - Colonoscopy, Lancaster, California
  - Advanced Imaging Center - Chest X-Ray, Lancaster, California
  - Antelope Valley Eye Care - Ophthalmologist, Lancaster, California
  - AV Pediatrics Allergy and Family Medicine, Lancaster, California
  - Jatinder S. Pruthi, MD FACG CPI, Lancaster, California
  - OM Research LLC, Lancaster, California
  - United Medical Doctors, Murrieta, California
  - Retina Consultants of Southern California, Victorville, California
  - Physicians Surgery Center, Victorville, California
  - Front Range Endoscopy Center, Colorado Springs, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Colorado Springs Pulmonary Consultants, PC, Colorado Springs, Colorado
  - The Wright Eye Center (OCT Facility), Colorado Springs, Colorado
  - Colorado Springs Imaging (Ultrasound and MRE Location), Colorado Springs, Colorado
  - Xera Med Research, Boca Raton, Florida
  - RecioMed Clinical Research Network, Inc, Boynton Beach, Florida
  - Florida Advanced Gastroenterology Center - Rahman Nakshabendi MD and Imad Nakshabendi, MD, Brandon, Florida
  - Bay Area Chest Physicians, P.A. (Pulmonary Function Test), Clearwater, Florida
  - West Coast Endoscopy Center (Endoscopy Procedures), Clearwater, Florida
  - Northwood Vision (Optical Coherence Tomography), Clearwater, Florida
  - Safety Harbor Surgery (Endoscopy Procedures), Clearwater, Florida
  - Gastro Florida (Regulatory Administrative Duties), Clearwater, Florida
  - Beraja Medical Institute (OCT), Coral Gables, Florida
  - Advanced Eye Center, Hialeah, Florida
  - UF Health Imaging Center-Emerson (chest x-rays), Jacksonville, Florida
  - UF Health Laboratory Emerson (blood draws), Jacksonville, Florida
  - UF Health Jacksonville Respiratory Therapy (PFT and DLCO), Jacksonville, Florida
  - UF Health Jacksonville-Faculty Clinic (ileocolonoscopy and biopsy), Jacksonville, Florida
  - UF Health Opthalmology - Jacksonville (Ophthalmology with OCT), Jacksonville, Florida
  - UF Health Radiology-Jacksonville (chest x-rays), Jacksonville, Florida
  - Cisca Pulmonary & Critical Care (PFT Facility), Jacksonville, Florida
  - Nicolitz Eye Consultants (OCT Facility), Jacksonville, Florida
  - Borland-Groover Clinic (Endoscopy Facility), Jacksonville, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Jupiter Outpatient Surgery Center, Jupiter, Florida
  - IHS Health, LLC, Kissimmee, Florida
  - Lee Shettle Eye & Hearing (Ophthalmoscopy Only), Largo, Florida
  - Infinite Clinical Research, Miami, Florida
  - Pulmonology Physicians of South Florida, Miami, Florida
  - Reina Eye Care P.A., Miami, Florida
  - The Endoscopy Center (Endoscopy Procedure), Miami, Florida
  - La Salud Research Clinic Inc., Miami, Florida
  - Research Associates of South Florida, Miami, Florida
  - South Florida Center for Endoscopy and Digestive Disease, LLC, Miami, Florida
  - Juan Barrio, MD (PFT when needed), Miami, Florida
  - Anchor Medical Research, Llc, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Gulfshore Endoscopy Center, Naples, Florida
  - Retina Consultants of Southwest Florida OCT only, Naples, Florida
  - Lisette Delgado Sanchez, MD PFT only, Naples, Florida
  - Pediatric & Adult Research Center, Orlando, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Bardmoor GastroEnterology, Seminole, Florida
  - Larkin Community Hospital (Endoscopy Procedure), South Miami, Florida
  - St. Petersburg Endoscopy Center (Endoscopy Procedures), St. Petersburg, Florida
  - Pasadena Center for Asthma and Lung Disorders (PFT and DLCO Only), St. Petersburg, Florida
  - Bay Area Endoscopy and Surgery Center (Endoscopy only), St. Petersburg, Florida
  - Theia Clinical Research, LLC, St. Petersburg, Florida
  - Advanced Research Institute Inc.(IP and PFT), St. Petersburg, Florida
  - Absolute Surgical Specialist - Craig Amshel, MD, Sun City Center, Florida
  - Lab - Processing/ Storage, Tampa, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - GCP Clinical Research,LLC, Tampa, Florida
  - LoCicero Medical Group, Tampa, Florida
  - Newsome Eye Specialist (OCT Procedures Only), Tampa, Florida
  - South Tampa Surgery Center, Tampa, Florida
  - USF Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Peachtree Allergy and Asthma Clinic - Chest X-rays and PFTs, Atlanta, Georgia
  - Ross Eyecare - Opthalmoscopy and OCT, Atlanta, Georgia
  - Atlanta Gastroenterology Associates (endoscopy only), Atlanta, Georgia
  - Atlanta Gastroenterology Associates(IP only), Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - GI Alliance, Arlington Heights, Illinois
  - Northwest Endoscopy Center (Endoscopy), Arlington Heights, Illinois
  - GI Alliance (PFT), Gurnee, Illinois
  - Illinois Gastroenterology Group-Gurnee (Patients Seen; IP Delivered), Gurnee, Illinois
  - Medical Eye Services LTD (Ophthalmoscopy with OCT), Gurnee, Illinois
  - North Shore Endoscopy Center (Endoscopy), Lake Bluff, Illinois
  - Libertyville Imaging Center (Diagnostic Imaging), Libertyville, Illinois
  - 3T Imaging of Morton Grove (Diagnostic Imaging), Morton Grove, Illinois
  - Charter Radiology, Columbia, Maryland
  - Cascades Endoscopy Center, Columbia, Maryland
  - Gastro Center of Maryland, LLC, Columbia, Maryland
  - Kaylani Eye Care ( Optical Coherence Tomography and Opthalmoscopy only), Hanover, Maryland
  - Lung Center (Pulmonary Function Test only), Laurel, Maryland
  - A Terrell Williams, MD, PLLC (OCT), Jackson, Mississippi
  - Jackson Pulmonary Associates (PFT), Jackson, Mississippi
  - Southern Therapy and Advanced Research, LLC, Jackson, Mississippi
  - St. Dominic Ambulatory Surgery Center (colonoscopy, Endoscopy), Jackson, Mississippi
  - Barnes-Jewish West County Hospital (Additional Endoscopy Location), Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Allied Health Clinical Research Organization, LLC, Freehold, New Jersey
  - Freehold Endoscopy Associates, LLC d/b/a Endoscopy Center of Monmouth County, Freehold, New Jersey
  - Freehold Ophthalmology, Freehold, New Jersey
  - Monmouth Ocean Pulmonary Medicine, Freehold, New Jersey
  - Princeton Radiology, Freehold, New Jersey
  - NYU Langone Eye Center (Ophthalmology), New York, New York
  - NYU Langone Health - Ambulatory Care Center, New York, New York
  - NYU Langone Health, Investigational Pharmacy, Perlmutter Cancer Center, New York, New York
  - NYU Langone Health, New York, New York
  - NYU Langone Inflammatory Bowel Disease Center, New York, New York
  - NYU Pulmonary and Critical Care Associates (Pulmonary), New York, New York
  - Queen City Gastroenterology and Hepatology (Endoscopy), Charlotte, North Carolina
  - Greenman Eye Associates (OCT), Charlotte, North Carolina
  - Carolinas Research Center, Charlotte, North Carolina
  - Cornerstone Medical (Imaging & PFT), Charlotte, North Carolina
  - Geauga Sleep Center(PFT only), Chardon, Ohio
  - UC Health Hoxworth (OCT only), Cincinnati, Ohio
  - UC Health Physicians Office, Cincinnati, Ohio
  - University of Cincinnati Medical Center (PFT and Endoscopy location), Cincinnati, Ohio
  - UC Health (Pulmonary Function Testing), Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Ophthalmic Physicians Incorporated (OCT Only), Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Vitreo Retinal Consultants(OCT only), Mentor, Ohio
  - Lake Pulmonary Associates (PFT only), Willoughby, Ohio
  - Retina Specialists of Ohio(OCT only), Willoughby Hills, Ohio
  - Norman Endoscopy Center, Norman, Oklahoma
  - Physicians and Surgeons X-Ray, Norman, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Saint Anthony Endoscopy Center, Oklahoma City, Oklahoma
  - SSM Health, Saint Anthony Hospital, Oklahoma City, Oklahoma
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Johnston Opthalmology, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - Houston Pulmonary Sleep and Allergy Associates (PFT), Cypress, Texas
  - Houston Eye Associates (For Eye Examination), Houston, Texas
  - Alkek Eye Center Jamail Specialty Care Center (OCT), Houston, Texas
  - Baylor College of Medicine - Baylor St. Luke's Medical Center, Houston, Texas
  - Baylor St. Luke's Medical Center - McNair Campus (pharmacy), Houston, Texas
  - Baylor St. Luke's Medical Center - McNair Campus, Houston, Texas
  - Baylor St. Luke's Medical Center Endoscopy - McNair Campus, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Mann Eye Institute, Houston, Texas
  - Memorial Hermann Hospital- TMC Investigational Drugs Services Pharmacy (Drug Storage), Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Bay Area Endoscopy Center, LLC, Houston, Texas
  - Pearland Surgery Center, Houston, Texas
  - Memorial Endoscopy Center (For Colonoscopy), Houston, Texas
  - Eye Specialists of Texas, Houston, Texas
  - Northside Gastroenterology Associates PA, Houston, Texas
  - Memorial Pulmonology(For PFT), Houston, Texas
  - Digestive Health Associates, Houston, Texas
  - Memorial Hermann Memorial City Digestive Health Center (For Colonoscopy), Houston, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Christus Trinity Mother Frances Endoscopy Center (endoscopies only), Tyler, Texas
  - Heaton Eye Associates (OCT only), Tyler, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - UT Health East Texas Physicians (pulmonary functions only), Tyler, Texas
  - Citizens Healthplex (for PFT only), Victoria, Texas
  - Surgery Center (For endoscopy only), Victoria, Texas
  - Victoria Eye Center (For OCT only), Victoria, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - GI Alliance Webster, Webster, Texas
  - Harman Eye Center (OCT only), Forest, Virginia
  - Lynchburg Pulmonary Associates, Inc. (PFT only), Lynchburg, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Swedish Endoscopy Center - Issaquah, Issaquah, Washington
  - Pacific Northwest Retina, Seattle, Washington
  - Richard Bensinger, MD, Seattle, Washington
  - Swedish Gastroenterology, Seattle, Washington
  - First Hill Endoscopy Center, Seattle, Washington
  - Pulmonary Function Lab, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Argentina (9):
  - Instituto Medico Elsa Perez(I.M.E.P), Ciudadela, Prov. de Buenos Aires
  - Instituto Medico Elsa Perez (I.M.E.P.) (Local Lab), Ciudadela, Prov. de Buenos Aires
  - Instituto Medico Elsa Perez (I.M.E.P.) (Pharmacy), Ciudadela, Prov. de Buenos Aires
  - Estudio de La Vision (OCT, Ophthalmoscopy), Hurlingham, Prov. de Buenos Aires
  - Gastroenterologia Rosario (Endoscopy), Rosario, Santa Fe Province
  - Microcirugia Ocular SA (OCT, Ophthalmoscopy), Rosario, Santa Fe Province
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Consultorios extemos de Sanatorio Parque (PFT with DLCO, Pulmonar Functional Test with DLCO), Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
- Australia (17):
  - Macquarie Respiratory Services, Macquarie University, New South Wales
  - Macquarie University Hospital Clinical Trials, Macquarie University, New South Wales
  - Macquarie University Hospital Pharmacy, Macquarie University, New South Wales
  - Macquarie University Hospital, Macquarie University, New South Wales
  - MQ Health Ophthalmology, Macquarie University, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - MCES Practice Pty Ltd operating as Comprehensive Eye Surgeons, Bellfield, Victoria
  - The Northern Hospital, Epping, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Footscray Hospital, Melbourne, Victoria
  - Vision Eye Institute, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Heidelberg Eye Clinic, Rosanna, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Lions Eye Institute Limited, Nedlands, Western Australia
  - The trustee for The RTS Unit Trust trading as Respiratory Testing Services, O'Connor, Western Australia
- Austria (5):
  - LKH Universitats-Klinikum Graz, Graz
  - Medical University Innsbruck, Internal Medicine Ⅰ, Innsbruck
  - AKH Wien- Universitatsklinik fiir Innere Medizin III, Vienna
  - AKH Wien- Universitatsklinik fur Innere Medizin III, Vienna
  - Univ.-Professor Dr. Mehrdad Baghestanian, Vienna
- Belarus (5):
  - Institution "Gomel Regional Clinical Hospital", Homyel
  - Health care Institution "10th City Clinical Hospital", Minsk
  - Health Care Institution "Mogilev Hospital #1", Mogilev
  - Health Care Institution "Vitebsk Regional Clinical Hospital", Vitebsk
  - Healthcare Institution "Vitebsk Regional Clinical Specialized Center", Vitebsk
- Belgium (7):
  - AZ Maria-Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - Campus Brugsesteenweg, Roeselare
  - Campus Rumbeke, Roeselare
  - Campus Rembert Torhout, Torhout
  - Centre Hospitalier Universitaire UCL Namur - Site Godinne, Yvoir
- Bulgaria (3):
  - "DCC Alexandrovska", EOOD, Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL" EAD, Sofia
  - ,,University multiprofile hospital for active treatment and emergency medicine N.I. Pirogov" EAD, Sofia
- Canada (7):
  - McGill University Health Centre - Montreal General Hospital (Electrocardiogram Clinic), Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital (Endoscopy Clinic), Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital (Pharmacy), Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital (Radiology), Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital (Research Site), Montreal, Quebec
  - Centre for Innovative Medicine - Research Institute of the McGill University Health Centre(Pulmonary, Montreal, Quebec
  - Eye Health MD (Ophthalmology), Montreal, Quebec
- Chile (3):
  - Centro de Investigaciones Clinicas de la Universidad Catolica, Santiago, RM
  - Clinica Universidad de los Andes, Santiago, Santiago Metropolitan
  - CeCim Biocinetic, Santiago, Santiago Metropolitan
- Colombia (4):
  - Clinica de la Costa Ltda., Barranquilla, Atlántico
  - Clinica de la Mujer S.A.S, Bogotá, Bogota D.C.
  - IPS Fundacion Cardiomet CEQUIN, Armenia, Quindío Department
  - Centro de lnvestigaciones Clinicas S.A.S, Cali, Valle del Cauca Department
- Croatia (2):
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital Center Zagreb, Zagreb
- Czechia (8):
  - MUDr. Jaroslava Skalova, Horažďovice
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - VISUS, spol s.r.o., Hradec Králové
  - GASTRO JeKa, s.r.o., Klatovy
  - Klatovska nemocnice a.s., Klatovy
  - MUDr. Pavlina Kazinotova s.r.o., Olomouc
  - Ocni ordinace Olomouc, Olomouc
  - PreventaMed s.r.o., Olomouc
- Denmark (2):
  - Aalborg University Hospital, Department of Medical Gastroenterology, Medicinerhuset, Aalborg
  - Hvidovre University Hospital, Hvidovre
- Egypt (8):
  - Alexandria Clinical Research Center , Faculty of Medicine , Alexandria University, Alexandria
  - Ain Shams University Hospital, Cairo
  - Air Force Specialized Hospital(AFSH), Cairo
  - Cairo University , Kasr Al Aini Hospital, Cairo
  - National Hepatology and Tropical Medicine Research Institute, Cairo
  - Egyptian Liver Research Institute and Hospital ( ELRIAH), Dakahlia
  - Theodor Bilharz Research Institute Research Ethics Committee, Giza
  - National Liver Institute, Menofeya
- France (21):
  - CHU Amiens Picardie, Amiens
  - CHU de Clermont Ferrand - Hopital Estaing, Clermont-Ferrand
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU Grenoble Alpes - Hopital Michallon, Grenoble
  - Endoscopy: CHU Grenoble Alpes- Hopital Michallon, Grenoble
  - CHD Vendee, Unite de Recherche Clinique, La Roche-sur-Yon
  - CHU de Lille - Hopital Claude Huriez, Lille
  - Optical Coherence Tomography and Ophthalmology CHU de Lille Hopital Roger Salengro, Lille
  - Pulmonary Function Test CHU Lille, Institut Coeur Poumon, Lille
  - CHU Saint-Eloi, Montpellier
  - Hopital Saint-Eloi - Pole Digestif - Hgea Recherche Clinique - Rdc, Montpellier
  - CHU de Nice, Hopital 1'Archet 2, Nice
  - Hopital Robert Debre, Reims
  - Hopital Maison Blanche, CHU DE REIMS, Reims
  - Hopital Robert Debre CHU DE REIMS, Reims
  - CHU Saint Etienne - Hopital Nord, Saint-Etienne
  - Optical Coherence Tomography and Ophthalmology, Saint-Priest-en-Jarez
  - Pulmonary Function Test, Saint-Priest-en-Jarez
  - Hopital Rangueil, Toulouse
  - Hopital Purpan PPR pole cephalique, Toulouse
  - Chru Nancy Brabois, Vandœuvre-lès-Nancy
- Georgia (7):
  - LLC 'Vivamedi', Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Academician Nikoloz Kipshidze Central University Clinic, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, LTD, Tbilisi
  - LTD Medical Center "CITO", Tbilisi
- Germany (16):
  - Gastroenterologie Opernstraβe, Kassel, Hassen
  - Universitaetsklinikum Augsburg, Augsburg
  - Staedtisches Klinikum Brandenburg, Brandenburg
  - Prof. Dr. med. Dr. med. Habil. Jens Buhren, FEBO, Frankfurt
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - HaFCED e.K. - Hamburgisches Forschungsinstitut für chronisch entzündliche Darmerkrankungen, Hamburg
  - OCT/Ophtalmoscopy address: Universitaetsklinikum Jena, Jena
  - PFT address: Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Jena, Jena
  - PFT address: Praxis fur Pneumologie und Allergologie, Kassel
  - OCT/Ophtalmoscopy address: Augenarztpraxis Dr. Karola Hassan, Kassel
  - Nordblick Augenklinik, Kiel
  - Universitatsklinikum Schleswig-Holstein- Campus Kiel, Kiel
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Dr. Irina Hasewinkel, Nürtingen
  - Medius Klinik Nuertingen, Nürtingen
- Greece (3):
  - Univerisity General Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Alexandroupoli, Alexandroupoli
  - General Hospital of Athens "Evangelismos", Athens
- Hungary (11):
  - Bugat Pal Korhaz, Gasztroenterologia, Gyöngyös, Heves County
  - DLCO and ophthalmology tests: Szent Borbala Korhaz, Tatabánya, Komárom-Esztergom
  - Szent Borbala Korhaz, Tatabánya, Komárom-Esztergom
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz, 4. Belgyogyaszat es 2. Gasztroenterologia, Békéscsaba
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft. (abbreviated name: Clinexpert Kft.), Budapest
  - Ophthalmology procedures: Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Pulmonary procedures: Vasutegeszsegugyi Nonprofit Kozhasznu K ft., Budapest
  - Semmelweis Egyetem, Belgyogyaszati es Hematologiai Klinika, Budapest
  - Ophthalmology, OCT: Medicover Zrt., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Chest X-ray: XIII. keruleti Egeszsegugyi Szolgalat Kozhasznu Nonprofit Kft., Budapest
- India (5):
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Fortis Memorial Research Institute, Gurugram, Haryana
  - Midas Multispeciality Hospital Pvt. Ltd, Nagpur, Maharashtra
  - S. R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Aster Medcity, Aster DM Healthcare Ltd., Kochi
- Israel (4):
  - HaEmek Medical Center, Afula
  - Shaare Zedek Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (16):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - OCT/ PFT/ Endoscopy address: IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - IRCCS Humanitas Research Hospital, Rozzano, Milano
  - ASST Rhodense - Pneumology Unit, Garbagnate Milanese, Milan
  - ASST Rhodense, U.O.C. Gastroenterologia ed Endoscopia Digestiva, Milan, Milan
  - ASST Rhodense - Ophthalmology Unit, Rho, Milan
  - Ospedale San Raffaele, Milan, MI
  - OCT/ PFT/ Endoscopy address: IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera Ospedale Cannizzaro, Catania
  - A.O. Mater Domini, U.O. Fisiopatologia Apparato Digerente Campus Universitario "Salvatore Venuta", Catanzaro
  - A.O. Mater Domini, U.O. Fisiopatologia Apparato Digerente, Catanzaro
  - CAMPUS GERMANETO Magazzino farmaci e dispositivi medici, uffici, Catanzaro
  - Fondazione IRCCS Policlinico San Matteo - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche, Pavia
  - PFT address: Azienda Ospedaliero-Universitaria Sant' Andrea UOC Pneumologia, Rome
  - IRCCS Ospedale Sacro Cuore Don Calabria, Verona
  - OCT/PFT/Endoscopy address: CRC - Cenro Ricerche Cliniche di Verona, Verona
- Japan (12):
  - Kokikai Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Ishii Eye Clinic, Nagareyama-shi, Chiba
  - Hospital of the university of occupational and environmental health, Kitakyushu-shi, Fukuoka
  - Kitakyushu Municipal Medical Center, Kitakyusyu-shi, Fukuoka
  - Matsumoto Eye Clinic, Toride-shi, Ibaraki
  - Kagoshima Kouseiren Hospital, Kagoshima, Kagoshima-ken
  - Jiaikai Idzuro Imamura Hospital, Kagoshima, Kagoshima-ken
  - Sameshima Eye Clinic, Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Saga University Hospital, Saga, Saga-ken
  - Japan Community Health care Organization Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
- Lebanon (5):
  - Saint George University Hospital Medical Center, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Hotel Dieu de France Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
  - Nini Hospital s.a:l, Tripoli
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Mexico (12):
  - Centro de Investigacion Medico Biologica Y Terapia Avanzada S.C., Guadalajara, Jalisco
  - Global Glaucoma Institute, Guadalajara, Jalisco
  - Video Endoscopia Americas, Guadalajara, Jalisco
  - Comercializadora Winco S.A. de C.V., Guadalajara, Jalisco
  - Cirugia y Gastro de Veracruz S.A. de C.V. (Progastro), Boca del Rio, Veracruz
  - Sanatorio Palmore A.C., Chihuahua City
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Vista Lasser de Chihuahua S.C., Chihuahua City
  - Servicios Hospitalarios de México, S.A. de C.V., Chihuahua City
  - FAICIC S. de R.L. de C.V., Veracruz
  - Gabinete de Diagnostico COVADONGA, Veracruz
  - Alberto Collado Solorzano (Clinica Vision), Veracruz
- Moldova (4):
  - "Sf. Arhanghel Mihail" Municipal Clinical Hospital, Department of Gastroenterology, Chisinau
  - PMSI Republican Clinical Hospital "Timofei Mosneaga", Department of Colorectal Surgery, Chisinau
  - PMSI Republican Clinical Hospital "Timofei Mosneaga", Department of Gastroenterology, Chisinau
  - PMSI Republican Clinical Hospital "Timofei Mosneaga", Outpatient Department, Chisinau
- Netherlands (2):
  - Academic Medical Centre, Amsterdam
  - UMC Utrecht, Utrecht
- Poland (36):
  - NSZOZ Termedica, Poznan, Greater Poland Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej (DLCO), Bystra
  - Specjalistyczne Gabinety Lekarskie LANDA, Karkow
  - Centre De La Vision Centrum Okulistyczne(OCT, Ophthalmoscopy), Krakow
  - Medicina (Endoscopy), Krakow
  - Centrum Medyczne EVITA(Endoscopy), Krakow
  - (Centrum Medyczne Ksiezy Mlyn (OCT and Ophthalmoscopy), Lodz
  - Centrum Medyczne "Ksiezy Mlyn" (OCT, Ophtalmoscopy), Lodz
  - AMICARE Sp. z o.o. sp.k, Lodz
  - IP Clinic Sp. z o.o., Lodz
  - Centra Medyczne Medyceusz (DLCO), Lodz
  - Salve Health Care Sp. o.o., (PFT and Endoscopy), Lodz
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatolog i im. M. Kopernika w Lodzi, Lodz
  - Allmedica Badania Kliniczne Sp. z o.o. Sp. k., Nowy Targ
  - Medicome Sp. Z O.O, Oświęcim
  - Przychodnia Okulistyczna "Oculus" Barbara Cybulska (OCT, Ophtalmoscopy), Piotrkow Trybunalski
  - Samodzielny Szpital Wojewodzki im. Mikolaja Kopernika (Endoscopy), Piotrkow Trybunalski
  - Trialmed CRS, Piotrokow Trybunalski
  - Solurmed Centrum Medyczne, Poznan
  - OCU Service Mikolaj Meller Sp.j.(OCT, Ophtalmoscopy), Poznan
  - Kliniczny Szpital Wojewodzki Nr 1 im. Fryderyka Chopina w Rzeszowie (Ophthalmpscopy), Rzeszów
  - Podkarpackie Centrum Chorob Plue w Rzeszowie (DLCO), Rzeszów
  - Centrum Medyczne Medyk, Rzeszów
  - Strzegomskie Centrum Medyczno - Diagnostyczne Sp. z o.o. (Endoscopy), Strzegom
  - Centrum Medyczne EZ-MEDICA (OCT, Ophtalmoscopy), Swidnica
  - DC-MED, Swidnica
  - Szpital "Latawiec" -Poradnia Gruzlicy i Chorob Pluc (PFT), Swidnica
  - Centrum Zdrowia MDM (OCT,opthalmoscopy), Warsaw
  - Centrum Zdrowia MDM, Warsaw
  - Instytut Gruzlicy i Chorob Pluc(DLCO), Warsaw
  - Endoterapia PFG (Endoscopy), Warsaw
  - Instytut Oka (OCT, Ophtalmoscopy), Warsaw
  - Specjalistyczne Gabinety Lekarskie Body Clinic, Warsaw
  - Centrum Okulistyczne JASKRA (OCT, Ophthalmoscopy), Warsaw
  - Wojskowy lnstytut Medyczny (PFT), Warsaw
  - EuroMediCare Szpital Specjalistyczny z Przychodniit (Endoscopy), Wroclaw
- Romania (4):
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca, JUD. CLUJ
  - Centrul de Diagnostic si Tratament Affidea, Specialitatea Medicina Interna, Constanța, Jud.constanta
  - SC Centrul Medical Medicum SRL, Specialitatea Gastroenterologie, Bucharest
  - Institutul Clinic Fundeni, Centrul de Gastroenterologie si Hepatologie, Bucharest
- Russia (14):
  - LLC "Polyclinic of ultrasonography 4D", Pyatigorsk, Stavropol Kray
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - LLC "SibNovoMed", Novosibirsk
  - Gastrocenter, Novosibirsk
  - LLC "Novosibirskiy Gastrocentr'', Novosibirsk
  - Hospital #12, Novosibirsk
  - LLC "Siberian Center for Prevention and Treatment of Myopia Eye", Novosibirsk
  - Joint Stock Company Medical Center "AVICENNA", Novosibirsk
  - BHI of Omsk region "Clinical oncology dispensary", Omsk
  - Clinicodiagnostic Center "Ultramed", Omsk
  - Medical center "Intervzglyad", Omsk
  - FSBI of Higher Education " North-Western Medical University n.a.I.I. Mechnikov '' of MoH RF, Saint Petersburg
  - FSBI of Higher Education "North-Western Medical University n.a.I.I. Mechnikov'' of MoH RF, Saint Petersburg
  - Autonomous Noncommercial Medical Organization "Stavropol Regional Clinical, Stavropol
- Clinical Center Zvezdara, Belgrade, Serbia
- Slovakia (9):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta, Banská Bystrica
  - ALIAN. s.r.o .. Ambulancia vnutorneho lekarstva, Bardejov
  - ENDOMED, s.r.o. Gastroenterologicka ambulancia, Košice
  - Opthalmology outpatient clinic, MUDr. Michal Popovec, s.r.o., Lipany
  - KM Management spol.s.r.o. Gastroenterologicke a hepatologicke centrum, Nitra
  - GASTRO I., s.r.o. Gastroenterologicka ambulancia, Prešov
  - GASTRO LM s.r.o., Gastroenterologicka ambulancia, Prešov
  - Pneumology: PULMO, s.r.o., Prešov
  - X-ray: FNsP J.A. Reimana Presov, Prešov
- South Africa (21):
  - Dr W Simmonds (Gastroenterology Department), Bloemfontein, Free State
  - Dr K Rahman (OTC and Opthalmoscopy), Benoni, Gauteng
  - Lakeview Hospital radiology (Radiology), Benoni, Gauteng
  - Worthwhile Clinical trials (PFT), Benoni, Gauteng
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Dr E Meyer & Partners, Centurion Eye Hospital (OTC and Opthalmoscopy), Centurion, Gauteng
  - Dr Jorg Reichenberger (Endoscopy), Centurion, Gauteng
  - Drs Burger Radiologists Inc (X-ray/CT), Centurion, Gauteng
  - Johese Clinical Research, Unitas Hospital, Centurion, Gauteng
  - WITS Clinical Research, Johannesburg, Gauteng
  - Burger Radiology (Radiology), Kempton Park, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Dr KJP Lubuya (OCT and Opthalmology), Kempton Park, Gauteng
  - Prof O Mwantembe (Endoscopy), Kempton Park, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - Dr K Rahman(OTC and Opthalmoscopy), Springs, Gauteng
  - Dr I Moola (Endoscopy), Sunninghill, Gauteng
  - Dr Peter Chapman (PFT + DLCO), Cape Town, Western Cape
  - Dr Chris Stander (OCT), Cape Town, Western Cape
  - Morton & Partners Radiologists (Radiology), Cape Town, Western Cape
  - Spoke Research Inc. Room 109, Cape Town, Western Cape
- South Korea (12):
  - DongGuk University ilsan Hospital, Goyang-si, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Endoscopy Facility in kyungpook National University Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - OCT Facility In kyungpook National University Hospital, Daegu
  - PFT Facility in Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon
  - Gachon university Gil Medical Center, Incheon
  - CHA University Bundang CHA Hospital, Seongnam-si
  - Kyunghee University Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (3):
  - Hospital General de Tomelloso, Tomellso, Ciudad REAL
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
- Switzerland (2):
  - Inselspital Bern, Bern
  - OCT/Ophtalmoscopy: Berner Augenklinik am Lindenhofspital, Bern
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - T.C. Saglik Bakanligi Ankara Sehir Hastanesi, Ankara
  - Saglik Bilimleri Universitesi Antalya Egitim ve Arastirma Hastanesi, Antalya
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Kocaeli University Research and Training Hospital, Kocaeli
  - Mersin University Faculty of Medicine, Yenişehir
- Ukraine (14):
  - Llc "Ldts Skaymed', Kharkiv
  - LLC "EyeQClinic", Kharkiv
  - Communal Non-commercial Enterprise Prof. O.O. Shalimov City Clinical Hospital #2 of Kharkiv, Kharkiv
  - Llc "Medical Center Oftalmika", Kharkiv
  - Municipal Health Care "Kharkiv City Hospital Ambulance and Emergency Medical care, Kharkiv
  - Communal Non-commercial Enterprise City Clinical Hospital #13 of Kharkiv City Council, Kharkiv
  - Medical Center of Limited Liability Company Harmoniia Krasy, Kyiv
  - Med Center 'Ok!Clinic+' of Comp with limited liability "Int Inst of Clin Research", Unit of Gastro, Kyiv
  - Private Enterprise "Clinic Medicom", Kyiv
  - CE Volyn Reg Clinical Hospital ofVolyn Reg Council, Surgical (Endocrine and Abdominal Pathology), Lutsk
  - Private Enterprise Diagnostic Center "Mediscan", Vinnytsia
  - Medical Center of LLC Health Clinic, Medical Clinical Research Center, Unit of Gastroenterology,, Vinnytsia
  - CNE of M.I. Pyrohov Vinnytsia Regional Clinical Hospital of Vinnytsia Regional Council, Reg, Vinnytsia
  - Scientific and Research Institute of Invalid Rehabilitation (Educational, Scientific and Treatment, Vinnytsia
- United Kingdom (4):
  - Royal Liverpool University Hospital, Liverpool
  - Central Middlesex Hospital, London
  - Guys & St Thomas Hospital, London
  - Quadram Institute Clinical Research Facility, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Dubinsky MC, Wu J, McDonnell A, Lazin K, Goetsch M, Branquinho D, Modesto I, Armuzzi A. Low Incidence of Macular Edema and Other Ocular Events in the Etrasimod Development Program. J Crohns Colitis. 2025 May 8;19(5):jjae173. doi: 10.1093/ecco-jcc/jjae173. PMID 39575597
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-202